CLINICAL TRIAL: NCT00770523
Title: Unrelated Donor Hematopoietic Stem Cell Transplantation After Nonmyeloablative Conditioning for Younger Patients With Hematologic Malignancies
Brief Title: Conditioning Regimen Before Infusion of Allogeneic Hematopoietic Stem Cells
Status: Completed | Type: Observational
Sponsor: Cooperative Study Group A for Hematology (Network)
Responsible Party: Yae-Eun Jang, COSAH
Other Study IDs: C-004
Record Dates: First submitted 2008-10-05; First posted 2008-10-10 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: HEMATOLOGIC MALIGNANCIES
Keywords: patients without comorbidity
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Unrelated Donor Hematopoietic Stem Cell Transplantation After Nonmyeloablative Conditioning for Younger Patients with Hematologic Malignancies.

DETAILED DESCRIPTION:
Primary end points are treatment-related mortality and engraftment. Secondary end points are regimen-related toxicities, graft-versus-host-disease, relapse, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

-Patients should have an unrelated donor who is matched for HLA-A and -B by serology and for -DRB1 by molecular typing.

Exclusion Criteria:

* Patients should not have major illness or organ failure
* Patients must not have a psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible.
* Patients must not be pregnant or lactating.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: acute leukemia chronic myelogenous leukemia myelodysplastic syndrome
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2003-12; Primary Completion 2008-03 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
treatment-related mortality and engraftment | all cause mortality

SECONDARY OUTCOMES:
regimen-related toxicities, graft-versus-host-disease, relapse, and overall survival. | Time point(s) at which outcome measure is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Kyoo-hyung Lee, doctor, Principal Investigator — COSAH
Locations (1):
- Asan Medical Center, Seoul, South Korea